CLINICAL TRIAL: NCT06754306
Title: A Randomized Controlled Trial on the Dynamic Effects of Different Dietary Interventions on Visceral Fat and Other Biochemical Markers
Brief Title: Dynamic Effects of Different Dietary Interventions on Visceral Fat and Biochemical Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: School of Public Health, Shanghai Jiao Tong University (Unknown); Huangpu District Center for Disease Control and Prevention, Shanghai (Unknown)
Responsible Party: Principal Investigator, Hui Wang, Principal Investigator, Professor, and Doctor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SJUPN-2024-009-HY1-KS2
Record Dates: First submitted 2024-12-18; First posted 2024-12-31 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Energy Metabolism
Keywords: Dietary Intervention; Randomized Controlled Trial; Intermittent Fasting; Caloric Restriction
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Balanced diet group (Experimental): Daily intake of 100% energy requirements, adjusted individually based on each participant's basal metabolic rate (BMR) and activity level.
  Interventions: Other: Balanced diet (100% energy)
- 16+8 time-restricted eating group (100% energy) (Experimental): Participants will consume 100% energy within an 8-hour eating window and fast for the remaining 16 hours.
  Interventions: Other: 16+8 time-restricted eating group (100% energy)
- 16+8 time-restricted eating group (75% energy) (Experimental): Participants will consume 75% of their energy requirements within the 8-hour eating window.
  Interventions: Other: 16+8 time-restricted eating group (75% energy)
- Alternate-day fasting group (75% energy) (Experimental): Participants alternate between "feeding days" (125% energy requirements) and "fasting days" (25% energy requirements).
  Interventions: Other: Alternate-day fasting group (75% energy)
- 5+2 intermittent fasting group (75% energy) (Experimental): Participants consume 95% energy requirements for 5 consecutive days and 25% energy requirements for 2 fasting days.
  Interventions: Other: 5+2 intermittent fasting group (75% energy)
- Low-calorie diet group (75% energy) (Experimental): Participants will reduce daily caloric intake to 75% of energy requirements, consumed evenly across three meals.
  Interventions: Other: Low-calorie diet group (75% energy)
- Very low-calorie diet group (45% energy) (Experimental): Participants will reduce daily caloric intake to 45% of energy requirements (~800 kcal/day)
  Interventions: Other: Very low-calorie diet group (45% energy)

INTERVENTIONS:
Other: Balanced diet (100% energy) — Daily intake of 100% energy requirements, adjusted individually based on each participant's basal metabolic rate (BMR) and activity level.
  Arms: Balanced diet group
Other: 16+8 time-restricted eating group (100% energy) — Participants will consume 100% energy within an 8-hour eating window and fast for the remaining 16 hours.
  Arms: 16+8 time-restricted eating group (100% energy)
Other: 16+8 time-restricted eating group (75% energy) — Participants will consume 75% of their energy requirements within the 8-hour eating window.
  Arms: 16+8 time-restricted eating group (75% energy)
Other: Alternate-day fasting group (75% energy) — Participants alternate between "feeding days" (125% energy requirements) and "fasting days" (25% energy requirements).
  Arms: Alternate-day fasting group (75% energy)
Other: 5+2 intermittent fasting group (75% energy) — Participants consume 95% energy requirements for 5 consecutive days and 25% energy requirements for 2 fasting days.
  Arms: 5+2 intermittent fasting group (75% energy)
Other: Low-calorie diet group (75% energy) — Participants will reduce daily caloric intake to 75% of energy requirements, consumed evenly across three meals.
  Arms: Low-calorie diet group (75% energy)
Other: Very low-calorie diet group (45% energy) — Participants will reduce daily caloric intake to 45% of energy requirements (~800 kcal/day)
  Arms: Very low-calorie diet group (45% energy)

SUMMARY:
This randomized clinical trial aims to evaluate the dynamic effects of various dietary interventions on visceral fat and biochemical markers among healthy adults. Participants aged 18-35 years with a normal body mass index (BMI 18.5-23.9) will be recruited from the community. Exclusion criteria include metabolic diseases, unstable weight, medication use, or pregnancy.

Participants will be randomly assigned to one of seven groups: 1) balanced diet (100% energy), 2) time-restricted eating (16+8, 100% energy), 3) time-restricted eating (16+8, 75% energy), 4) alternate-day fasting (75% energy), 5) 5+2 fasting (75% energy), 6) low-calorie diet (75% energy), and 7) very low-calorie diet (45% energy). The intervention consists of a 1-week baseline phase, a 4-week dietary intervention phase, and a 28-week recovery phase.

Primary outcomes include changes in visceral fat area, while secondary outcomes include body composition, cardiovascular health indicators (e.g., blood pressure, cholesterol), inflammation markers, and liver/kidney function. Biological samples (blood, urine, and feces) will be collected at multiple time points to facilitate multi-omics analyses, including proteomics, metabolomics, metagenomics, and DNA methylation.

The study aims to compare the short-term effects of different dietary interventions and explore underlying biological mechanisms. Findings will provide evidence for public health policies and dietary guidelines related to weight management and metabolic health.

DETAILED DESCRIPTION:
This study is a randomized clinical trial (RCT) designed to investigate the effects of different dietary interventions on visceral fat, body composition, and various biochemical indicators. The study will also incorporate multi-omics analyses to explore the dynamic biological mechanisms underlying these effects.

Study Background The increasing burden of obesity and chronic diseases has raised global concerns about effective dietary strategies. Recent dietary approaches, such as intermittent fasting (e.g., 16:8, alternate-day fasting, and 5:2 fasting) and continuous caloric restriction, have shown potential benefits in weight management and metabolic health. However, there is a lack of systematic comparisons between these dietary interventions and insufficient understanding of their dynamic biological effects.

This study aims to compare the short-term impacts of various dietary interventions and identify the biological mechanisms influencing visceral fat and metabolic changes. Multi-omics analyses will include proteomics, metabolomics, metagenomics, DNA methylation etc. to provide a comprehensive understanding of these effects.

Study Design

This RCT will recruit 84 healthy adults (12 participants per group), aged 18-35 years, with a normal BMI (18.5-23.9). Participants will be randomly assigned to one of seven groups:

Balanced diet group: Daily intake of 100% energy requirements, adjusted individually based on each participant's basal metabolic rate (BMR) and activity level.

16+8 time-restricted eating group (100% energy): Participants will consume 100% energy within an 8-hour eating window and fast for the remaining 16 hours.

16+8 time-restricted eating group (75% energy): Participants will consume 75% of their energy requirements within the 8-hour eating window.

Alternate-day fasting group: Participants alternate between "feeding days" (125% energy requirements) and "fasting days" (25% energy requirements).

5+2 intermittent fasting group: Participants consume 95% energy requirements for 5 consecutive days and 25% energy requirements for 2 fasting days.

Low-calorie diet group (75% energy): Participants will reduce daily caloric intake to 75% of energy requirements, consumed evenly across three meals.

Very low-calorie diet group (45% energy): Participants will reduce daily caloric intake to 45% of energy requirements (~800 kcal/day).

The study will span 33 weeks and include three phases:

Baseline phase (1 week): Participants consume their usual diet, and baseline measurements are taken.

Intervention phase (4 weeks): Participants adhere to their assigned dietary intervention.

Recovery phase (28 weeks): Participants return to their usual diet. Participants will be monitored closely throughout the study to ensure adherence to the intervention and the stability of other lifestyle factors (e.g., physical activity).

Outcome Measures Primary outcome: Changes in visceral fat area. Secondary outcomes: Changes in body composition (waist circumference, BMI, body fat percentage), cardiovascular indicators (e.g., blood pressure, cholesterol levels), inflammation markers (e.g., IL-6, IL-8), and liver/kidney function.

Biological samples (blood, urine, and feces) will be collected at baseline, weekly during the intervention phase, and at weeks 5, 8 and 32 of the recovery phase. Samples will be analyzed using multi-omics techniques, including proteomics, metabolomics, metagenomics, DNA methylation, etc. to identify dynamic biological changes associated with the dietary interventions.

Data Collection and Analysis Participants' data will include questionnaires, anthropometric measurements, biochemical tests, and multi-omics results. Blood samples, urine samples, and fecal samples (2 will be collected at each time point. Data will be analyzed to compare group differences in primary and secondary outcomes, with additional exploration of the underlying biological mechanisms through omics analyses.

Ethical Considerations The study has received ethical approval from the Institutional Review Board for Public Health and Nursing Research, Shanghai Jiao Tong University School of Medicine. Informed consent will be obtained from all participants before enrollment. Participant privacy and data confidentiality will be strictly maintained throughout the study.

Significance This study will provide a comparative analysis of different dietary interventions and their impacts on visceral fat and metabolic health. The inclusion of dynamic multi-omics analyses will offer new insights into the biological mechanisms underlying these effects. The findings will contribute valuable evidence for the development of dietary guidelines and public health strategies for weight management and chronic disease prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18-35 years.
2. BMI between 18.5 and 23.9.
3. Willing to voluntarily sign the informed consent form and comply with group assignments and intervention protocols.

Exclusion Criteria:

1. Diagnosed with metabolic diseases such as hypertension, diabetes, or dyslipidemia.
2. Diagnosed with uncontrolled psychiatric disorders.
3. Diagnosed with severe underlying diseases, such as renal failure, heart failure, or cancer.
4. Currently taking medications that may affect study outcomes (e.g., antihypertensive, antidiabetic, or lipid-lowering drugs).
5. Women in the perimenopausal stage or with irregular menstrual cycles.
6. Pregnant women.
7. Current smokers.
8. Unstable weight within the past three months (fluctuations exceeding 4 kg).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Change in Visceral Fat Area over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
  Visceral fat area will be measured using the InBody770 bioelectrical impedance analysis (BIA) device.

SECONDARY OUTCOMES:
Change in Body Weight over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
Change in Waist Circumference over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
Change in Hip Circumference over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
Body height at Baseline | Baseline only
Change in Body Mass Index (BMI) over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
  Body Weight and height will be used to calculate BMI in kg/m^2.
Change in Body Fat Mass over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
  Body fat mass will be measured using the InBody770 bioelectrical impedance analysis (BIA) device.
Change in Percent Body Fat Mass over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
  Percent body fat will be measured using the InBody770 bioelectrical impedance analysis (BIA) device.
Change in Skeletal Muscle Mass over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
  Skeletal muscle mass will be measured using the InBody770 bioelectrical impedance analysis (BIA) device.
Change in Visceral Fat Level over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
  Visceral fat level will be measured using the InBody770 bioelectrical impedance analysis (BIA) device.
Change in Basal Metabolic Rate over the Course of the Dietary Intervention | Baseline, and Week 4
  Basal metabolic rate will be measured using the metabolic cart.
Change in Blood Pressure over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
Change in Blood lipids over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
  Lipid profile measurements will include the following biomarkers: Apolipoprotein B (Apo-B), Lipoprotein(a) [LPa], Apolipoprotein A1 (Apo-A1), Low-Density Lipoprotein Cholesterol (LDL-C), High-Density Lipoprotein Cholesterol (HDL-C), Triglycerides (TG), and Total Cholesterol (Tch).
Change in Blood glucose over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
Change in Inflammation Markers over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
  Inflammatory biomarkers will be measured to assess participants' systemic inflammatory status and immune response. The panel of biomarkers includes interleukins (IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12p70, IL-17A), interferon-gamma (IFN-γ), tumor necrosis factors (TNF-α, TNF-β) and CRP.
Change in Liver Function Indicators over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
  Liver function will be assessed through blood biochemical analysis. Specific indicators include alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), albumin (ALB), total protein (TP), direct bilirubin (D-BIL), and total bilirubin (T-BIL).
Change in Kidney Function Indicators over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
  Kidney function will be assessed through blood biochemical analysis. Specific indicators include serum creatinine (SCr) and blood urea nitrogen (BUN).
Genetic Analysis Using ASA Chip | Baseline Only
Dynamic Changes in Multi-Omics Profiles (Methylation Chip, Blood Transcriptomics, Proteomics, Metabolomics, Fecal Metagenomics, and Fecal Metabolomics) over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
Changes in Urinalysis Indicators over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
  Urinalysis will be performed to assess general kidney function, metabolic status, and potential abnormalities in urinary composition. The panel of indicators includes leukocyte esterase, specific gravity, bilirubin, urobilinogen, protein, pH, glucose, ketones, nitrites, occult blood, and urine color.
Changes in Mental Health Status Measured by PHQ-9 over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
  The Patient Health Questionnaire-9 (PHQ-9) will be used to assess depressive symptoms. The PHQ-9 is a validated questionnaire with 9 items, scored on a scale from 0 to 3 for each item, resulting in a total score ranging from 0 to 27. Higher scores indicate worse mental health outcomes, with higher levels of depressive symptoms.
Changes in Mental Health Status Measured by SAS over the Course of the Dietary Intervention | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
  The Self-Rating Anxiety Scale (SAS) will be used to assess anxiety symptoms. The SAS consists of 20 items, with each item scored on a scale from 1 to 4, and the total raw score is converted to a standard score ranging from 25 to 100. Higher scores indicate worse mental health outcomes, with more severe anxiety symptoms.
Changes in Sleeping Status Measured by PSQI over the Course of the Dietary Intervention | Baseline, Week 4, Week 8, and Week 32
  The Pittsburgh Sleep Quality Index (PSQI) will be used to evaluate participants' sleep quality. The PSQI is a validated questionnaire with 19 self-rated items, generating 7 component scores (e.g., subjective sleep quality, sleep latency, sleep duration) that are combined into a global score. The global PSQI score ranges from 0 to 21, with higher scores indicating worse sleep quality.
Adverse Events Reporting over the Dietary Intervention Course | Week 1, Week 2, Week 3, Week 4, Week 5, Week 8, and Week 32
Continuous Glucose Monitoring Metrics over the Dietary Intervention Course | Continuously Throughout the Study (Baseline to Week 8)
  Dynamic tracking of glucose levels using a continuous glucose monitoring device to evaluate glycemic responses to dietary interventions.
Changes in Sleep Metrics Measured by Smart Ring over the Dietary Intervention Course | Continuously Throughout the Study (Baseline to Week 8)
  Sleep metrics, including duration, sleep stages, and overall sleep quality, will be continuously monitored using a smart ring. Measurements will provide insights into sleep patterns and changes over the study period.
Changes in Physical Activity Metrics Measured by Smart Ring over the Dietary Intervention Course | Continuously Throughout the Study (Baseline to Week 8)
  Physical activity metrics, including step count, activity duration, and intensity, will be continuously tracked using a smart ring to assess participants' activity levels throughout the study.
Changes in Blood Oxygen Levels (SpO₂) Measured by Smart Ring over the Dietary Intervention Course | Continuously Throughout the Study (Baseline to Week 8)
  Real-time blood oxygen saturation (SpO₂) will be continuously measured using a smart ring to monitor oxygen levels and detect any variations during the study.
Changes in Heart Rate Metrics Measured by Smart Ring over the Dietary Intervention Course | Continuously Throughout the Study (Baseline to Week 8)
  Heart rate metrics, including resting heart rate and activity-related heart rate, will be continuously monitored using a smart ring to assess cardiovascular response and changes over time.
Changes in Respiration Rate Measured by Smart Ring over the Dietary Intervention Course | Continuously Throughout the Study (Baseline to Week 8)
  Respiration rate will be continuously tracked using wearable devices, providing data on participants' breathing patterns and changes over the study period.
Changes in Stress Levels Measured by Smart Ring over the Dietary Intervention Course | Continuously Throughout the Study (Baseline to Week 8)
  Physiological stress indicators, such as heart rate variability (HRV) and other metrics, will be monitored using wearable devices to assess changes in participants' stress levels over the course of the study.
Changes in Blood Pressure Measured by Smart Watch over the Dietary Intervention Course | Continuously Throughout the Study (Baseline to Week 8)
  Blood pressure variations will be continuously measured using a smartwatch to monitor changes and trends in participants' cardiovascular health throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wang, PhD, Principal Investigator — School of Public Health, Shanghai Jiao Tong University School of Medicine, Shanghai, China
Locations (1):
- School of Public Health, Shanghai Jiao Tong University, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
We acknowledge the importance of data sharing for scientific advancement; however, due to the absence of a predefined data sharing mechanism in our study design and the need to prioritize participant confidentiality, we currently do not have a plan to share individual participant data (IPD). We remain open to exploring future opportunities to share aggregate data or collaborate with interested researchers within an ethically appropriate framework.